CLINICAL TRIAL: NCT02660554
Title: Rapid Diagnostic Testing to Guide Antibiotic Therapy in Drug Resistant Pneumonia
Brief Title: Trial of MRSA Polymerase Chain Reaction for Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Richard Wunderink, Professor, Department of Pulmonary and Critical Care Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STU00202148
Record Dates: First submitted 2016-01-04; First posted 2016-01-21 (Estimated); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Pneumonia; Methicillin-Resistant Staphylococcus Aureus
Keywords: Pneumonia; Methicillin-Resistant Staphylococcus aureus; Polymerase Chain Reaction; Intensive care units; Drug Resistance
MeSH Terms: conditions — Pneumonia | interventions — Polymerase Chain Reaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care (No Intervention): In the usual care arm, antibiotic therapy against methicillin resistant Staphylococcus aureus (MRSA) will be given at the discretion of the care team. If bacterial cultures are negative for MRSA at 72 hours, the treating physician will be prompted to discontinue MRSA therapy.
- Polymerase Chain Reaction (Experimental): In subjects randomized to the polymerase chain reaction (PCR) arm, antibiotic therapy against methicillin resistant Staphylococcus aureus (MRSA) will be determined by the results of the PCR test. In subjects who are clinically stable, results from the PCR must be available prior to the administration of MRSA therapy. Subjects with a positive MRSA PCR will be administered MRSA therapy. In subjects with a negative MRSA PCR, MRSA therapy will be withheld. In subjects randomized to the automated PCR arm who are clinically unstable, empiric MRSA therapy will be allowed until the PCR is completed. In these cases of unstable subjects, empiric MRSA therapy will be discontinued if the PCR is negative.
  Interventions: Other: Polymerase Chain Reaction (PCR)

INTERVENTIONS:
Other: Polymerase Chain Reaction (PCR) — Respiratory samples called bronchoalveolar lavage (BAL) gathered from subjects in the PCR arm will be tested for the presence of MRSA using the Cepheid Xpert® Assay. Xpert® is a qualitative in vitro test designed for rapid detection and differentiation of Staphylococcus aureus (SA) and methicillin resistant Staphylococcus aureus (MRSA) using PCR amplification. MRSA is identified by the mecA gene and staphylococcal cassette chromosome mec (SCCmec). Xpert® Assay is approved by the Federal Drug Administration to detect MRSA in soft tissue samples. Once the PCR is completed, the results will be relayed to the treating physician, and antibiotic therapy (vancomycin or linezolid) will be started or stopped based on the study protocol. All BAL samples will be sent for routine bacterial cultures.
  Arms: Polymerase Chain Reaction

SUMMARY:
The purpose of this study is to conduct a randomized clinical trial to compare an antibiotic strategy based on a novel diagnostic test, polymerase chain reaction (PCR) to usual care, in critically ill adults with pneumonia suspected to be caused by methicillin resistant staphylococcus aureus (MRSA). The investigators hypothesize that when automated PCR is used to guide antibiotic therapy, antibiotic exposure will be reduced in critically ill subjects with pneumonia.

DETAILED DESCRIPTION:
Bacterial resistance to antibiotics is a major problem in intensive care units (ICUs). The Centers for Disease Control (CDC) estimate drug resistant infections affect more than 2 million individuals nationwide and cause 23,000 deaths annually. In a recent executive order, the President of the United States called for improved antibiotic stewardship and the development of rapid diagnostic tests to identify antibiotic resistant infections. In ICU patients with pneumonia, guidelines advocate the routine use of broad spectrum antibiotics in most patients. In large part this is because diagnostic testing for pneumonia is too insensitive and too slow to inform decision making about appropriate antibiotics. Overuse of broad spectrum antibiotics promotes drug resistance by selecting for antibiotic resistant bacterial strains. This proposal will apply a new diagnostic test, polymerase chain reaction (PCR), to rapidly identify a drug resistant pathogen, methicillin resistant staphylococcus aureus (MRSA) to reduce inappropriate antibiotics in ICU patients with suspected pneumonia.

MRSA is an important cause of drug resistant pneumonia associated with high mortality. Methicillin resistance in Staphylococcus aureus (SA) results from acquisition of the mecA gene located in the mobile element staphylococcal cassette chromosome mec (SCCmec). MRSA pneumonia requires specific antibiotic therapy, treatment guidelines recommend addition of empiric antibiotics against MRSA in patients admitted to the ICU with risk factors for DRPs. The investigators prior work demonstrates that there is significant overlap of MRSA risk factors with risk factors for other DRPs, which potentially leads to the overuse of anti-MRSA antibiotics. Globally, MRSA pneumonia occurs in an estimated 2-6% of ICU patients. By contrast, empiric anti-MRSA therapy is prescribed in the majority of ICU patients with suspected pneumonia. The investigators have shown that at their own institution, the prevalence of MRSA is 5.5%, but empiric anti-MRSA therapy is prescribed in 89.5% of ICU patients with pneumonia. The large gap between empiric antibiotic therapy for MRSA pneumonia and actual cases of MRSA pneumonia is due to the lack of specificity of DRP risk factors, and the time delay of bacterial cultures. Overuse of antibiotics against MRSA has adverse consequences for patients, including new hospital acquired infections (HAIs), increased hospital length of stay (LOS), and higher cost.

Faster and more accurate diagnostic tests for MRSA, such as PCR, have the potential to reduce antibiotic exposure and improve patient outcomes. The time delay of bacterial cultures and the lack of specificity of DRP risk factors is a major limitation to the treatment of pneumonia, particularly in ICUs where the rapid delivery of appropriate antibiotics could be life saving. PCR has the potential to change the paradigm of empiric antibiotics by increasing diagnostic certainty and reducing the time to diagnosis or exclusion of a resistant pathogen. However, molecular diagnostic tests have not yet been validated for routine clinical practice.

The goal of this trial is to compare conduct a clinical trial to compare a PCR guided approach to MRSA therapy to usual care to determine if 1) an antibiotic strategy that utilizes rapid automated PCR reduces antibiotic-days in ICU subject with suspected pneumonia, 2) To compare the safety of an antibiotic strategy that relies on rapid automated PCR to usual care, and 3) To compare costs of the rapid automated PCR based strategy to routine microbiologic cultures.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 years and older with known or suspected pneumonia who are endotracheally intubated and mechanically ventilated
2. Can receive bronchoalveolar lavage (BAL) while intubated
3. Have received 24 hours or less of MRSA therapy (the antibiotics vancomycin or linezolid) prior to study enrollment

Exclusion Criteria:

1. More than 24 hours of MRSA therapy therapy (the antibiotics vancomycin or linezolid),
2. Subjects with extra pulmonary infection requiring treatment with vancomycin or linezolid
3. Neutropenic fever
4. Chronic airway infection
5. Patient/surrogate refusal
6. Subjects in whom BAL is deemed unsafe by the treating physician
7. Treating physician refusal to discontinue antibiotics to treat MRSA if PCR negative
8. Prisoners
9. Pregnant women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-01; Primary Completion 2017-02-28 (Actual); Study Completion 2019-05-03 (Actual)

PRIMARY OUTCOMES:
Days of anti-MRSA antibiotic therapy | 14 days
  days for initially suspected MRSA pneumonia

SECONDARY OUTCOMES:
Mortality | 28 days post randomization
  All cause mortality
Organ dysfunction | 28 days post randomization
  Days alive and organ dysfunction free for 28 days (based on daily SOFA score)
Renal Organ dysfunction | 28 days post randomization
  Days alive and renal organ dysfunction free for 28 days (based on daily SOFA renal organ score)
Days of subsequent anti-MRSA treatment | 28 days post randomization
  total days of vancomycin or linezolid treatment

CONTACTS AND LOCATIONS:
Overall Officials: Richard G Wunderink, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

REFERENCES:
- [Background] Wunderink RG. How important is methicillin-resistant Staphylococcus aureus as a cause of community-acquired pneumonia and what is best antimicrobial therapy? Infect Dis Clin North Am. 2013 Mar;27(1):177-88. doi: 10.1016/j.idc.2012.11.006. Epub 2012 Dec 14. PMID 23398873
- [Background] Shindo Y, Ito R, Kobayashi D, Ando M, Ichikawa M, Shiraki A, Goto Y, Fukui Y, Iwaki M, Okumura J, Yamaguchi I, Yagi T, Tanikawa Y, Sugino Y, Shindoh J, Ogasawara T, Nomura F, Saka H, Yamamoto M, Taniguchi H, Suzuki R, Saito H, Kawamura T, Hasegawa Y. Risk factors for drug-resistant pathogens in community-acquired and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2013 Oct 15;188(8):985-95. doi: 10.1164/rccm.201301-0079OC. PMID 23855620
- [Background] Kollef MH, Micek ST. Strategies to prevent antimicrobial resistance in the intensive care unit. Crit Care Med. 2005 Aug;33(8):1845-53. doi: 10.1097/01.ccm.0000171849.04952.79. PMID 16096464
- [Background] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079
- [Background] Mandell LA, Wunderink RG, Anzueto A, Bartlett JG, Campbell GD, Dean NC, Dowell SF, File TM Jr, Musher DM, Niederman MS, Torres A, Whitney CG; Infectious Diseases Society of America; American Thoracic Society. Infectious Diseases Society of America/American Thoracic Society consensus guidelines on the management of community-acquired pneumonia in adults. Clin Infect Dis. 2007 Mar 1;44 Suppl 2(Suppl 2):S27-72. doi: 10.1086/511159. No abstract available. PMID 17278083
- [Background] Haley CC, Mittal D, Laviolette A, Jannapureddy S, Parvez N, Haley RW. Methicillin-resistant Staphylococcus aureus infection or colonization present at hospital admission: multivariable risk factor screening to increase efficiency of surveillance culturing. J Clin Microbiol. 2007 Sep;45(9):3031-8. doi: 10.1128/JCM.00315-07. Epub 2007 Jul 11. PMID 17626171
- [Background] Rimawi RH, Mazer MA, Siraj DS, Gooch M, Cook PP. Impact of regular collaboration between infectious diseases and critical care practitioners on antimicrobial utilization and patient outcome. Crit Care Med. 2013 Sep;41(9):2099-107. doi: 10.1097/CCM.0b013e31828e9863. PMID 23873275
- [Background] Raman K, Nailor MD, Nicolau DP, Aslanzadeh J, Nadeau M, Kuti JL. Early antibiotic discontinuation in patients with clinically suspected ventilator-associated pneumonia and negative quantitative bronchoscopy cultures. Crit Care Med. 2013 Jul;41(7):1656-63. doi: 10.1097/CCM.0b013e318287f713. PMID 23528805
- [Background] Goff DA, Jankowski C, Tenover FC. Using rapid diagnostic tests to optimize antimicrobial selection in antimicrobial stewardship programs. Pharmacotherapy. 2012 Aug;32(8):677-87. doi: 10.1002/j.1875-9114.2012.01137.x. PMID 23307517
- [Background] Cercenado E, Marin M, Burillo A, Martin-Rabadan P, Rivera M, Bouza E. Rapid detection of Staphylococcus aureus in lower respiratory tract secretions from patients with suspected ventilator-associated pneumonia: evaluation of the Cepheid Xpert MRSA/SA SSTI assay. J Clin Microbiol. 2012 Dec;50(12):4095-7. doi: 10.1128/JCM.02409-12. Epub 2012 Sep 19. PMID 22993185
- [Background] Oh AC, Lee JK, Lee HN, Hong YJ, Chang YH, Hong SI, Kim DH. Clinical utility of the Xpert MRSA assay for early detection of methicillin-resistant Staphylococcus aureus. Mol Med Rep. 2013 Jan;7(1):11-5. doi: 10.3892/mmr.2012.1121. Epub 2012 Oct 9. PMID 23064681
- [Background] Leone M, Malavieille F, Papazian L, Meyssignac B, Cassir N, Textoris J, Antonini F, La Scola B, Martin C, Allaouchiche B, Hraiech S; AzuRea Network. Routine use of Staphylococcus aureus rapid diagnostic test in patients with suspected ventilator-associated pneumonia. Crit Care. 2013 Aug 6;17(4):R170. doi: 10.1186/cc12849. PMID 23919575
- [Background] Salgado CD, Farr BM, Calfee DP. Community-acquired methicillin-resistant Staphylococcus aureus: a meta-analysis of prevalence and risk factors. Clin Infect Dis. 2003 Jan 15;36(2):131-9. doi: 10.1086/345436. Epub 2003 Jan 3. PMID 12522744
- [Derived] Paonessa JR, Shah RD, Pickens CI, Lizza BD, Donnelly HK, Malczynski M, Qi C, Wunderink RG. Rapid Detection of Methicillin-Resistant Staphylococcus aureus in BAL: A Pilot Randomized Controlled Trial. Chest. 2019 May;155(5):999-1007. doi: 10.1016/j.chest.2019.02.007. Epub 2019 Feb 15. PMID 30776365

DOCUMENTS (1):
  • Study Protocol (2016-09-09): https://cdn.clinicaltrials.gov/large-docs/54/NCT02660554/Prot_000.pdf